CLINICAL TRIAL: NCT02520674
Title: Glaucoma Screening With Smartphone Ophthalmology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi di Brescia (Other)
Responsible Party: Principal Investigator, Andrea Russo, MD, PhD Candidate, Università degli Studi di Brescia
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: SMART002
Record Dates: First submitted 2015-08-03; First posted 2015-08-13 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Glaucoma and Ocular Hypertension (Other): Patients to be examined with both smartphone ophthalmoscopy and slit-lamp biomicroscopy.
  Interventions: Other: optic nerve head ophthalmoscopy

INTERVENTIONS:
Other: optic nerve head ophthalmoscopy — Patients underwent undilated smartphone ophthalmoscopy followed by undilated slit-lamp biomicroscopy for the grading of the vertical cup-to-disc ratio of the optic nerve head.

SUMMARY:
The purpose of this study is to assess the accuracy and reliability of smartphone ophthalmoscopy compared to slit-lamp biomicroscopy in glaucoma screening for potential community screening programs.

ELIGIBILITY:
Inclusion Criteria:

* ocular hypertension
* glaucoma

Exclusion Criteria:

* substantial media opacity
* refractive error outside the range from -10.00 to +5.00 diopters

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2014-09; Primary Completion 2015-06 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Vertical cup-to-disc ratio | Up to 25 weeks from date of study initiation